CLINICAL TRIAL: NCT06621784
Title: The Effect of Core Stabilization Exercises on Pain, Function, Balance, and Quadriceps Muscle Thickness in Patients with Knee Osteoarthritis
Brief Title: Core Stabilization Exercises in Patients with Knee Osteoarthritis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, İrem Setenay Özkan, Resident, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023/377
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-09

CONDITIONS: Exercise Training; Osteoarthritis, Knee; Core Stability; Muscle Thickness of the Quadriceps Femoris; Balance
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Traditional exercise (control) group (Active Comparator): The first group followed a standard home exercise program for three times per week for six weeks
  Interventions: Other: Classical exercise therapy
- core exercise group (Active Comparator): The second group followed a standard home exercise program and core stabilization exercises for three times per week for six weeks
  Interventions: Other: Core stabilization exercises; Other: Classical exercise therapy

INTERVENTIONS:
Other: Core stabilization exercises — In most studies, exercises focused on the extremities have been researched. We believe that the positive effects of the core region on walking and postural stability will play a significant role in the treatment of knee osteoarthritis.
  Arms: core exercise group
Other: Classical exercise therapy — In the first group of our study, we prescribed exercises that have been proven effective in many studies, are frequently prescribed, and focus on joint range of motion and quadriceps strengthening

SUMMARY:
Exercise plays a key role in the treatment of knee osteoarthritis, but there is no clear evidence on which type of exercise is most effective. Recent studies highlight the benefits of core stabilization exercises for improving knee stability. This study aims to demonstrate the effects of adding core stabilization exercises to conventional exercise therapy for patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Knee osteoarthritis is becoming a significant public health problem with the aging population. While there is no definitive cure, exercise is the main approach to treatment. Various types of exercises are being studied for their effectiveness in osteoarthritis treatment, and recently, core stabilization exercises have been highlighted for their role in lower extremity pathologies. In this study, we aimed to investigate the effects of these exercises on pain, balance, quality of life, function, and quadriceps muscle thickness in patients with knee osteoarthritis.

This study was designed as a randomized controlled double-blind clinical trial. Thirty-two patients were randomly divided into two groups: a conventional exercise group and a conventional+core group. A total of 18 home exercise sessions, performed three times per week for six weeks, were planned.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bilateral stage II or III knee osteoarthritis according to the Kellgren and Lawrence grading system
* Aged between 50 and 65 years
* Having a complaint of knee pain for at least 6 months
* No systemic diseases that may hinder exercise (such as uncontrolled hypertension, cardiac arrhythmia, heart failure, neurological sequelae, joint deformities, malignancy, etc.)

Exclusion Criteria:

* Having received physical therapy in the last 6 months
* Having undergone knee injection in the last 6 months
* Having had knee surgery
* Morbid obesity
* Presence or history of malignancy
* Individuals with severe visual impairment
* Individuals with a history of neurological or vestibular diseases that could cause balance problems, or patients using medications that may affect balance
* Individuals with serious cardiac, respiratory, or uncontrolled metabolic diseases

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-06-23 (Actual); Primary Completion 2024-06-23 (Actual); Study Completion 2024-10-09 (Estimated)

PRIMARY OUTCOMES:
Change in Knee Injury and Osteoarthritis Outcome Score total and subscale scores after a 6-week exercise program | Baseline and 1 week after the 6-week exercise program
  The Knee Injury and Osteoarthritis Outcome Score is scored on a scale from 0 to 100, where 0 represents extreme knee problems and 100 indicates no knee problems. Higher scores indicate a better outcome, reflecting less pain and better function.

SECONDARY OUTCOMES:
Change in single-leg stance test durations after a 6-week exercise program | Baseline and 1 week after the 6-week exercise program
  In the Single Leg Stance Test, the participant is initially asked to keep their eyes open. Then, one foot is lifted without touching the supporting leg. The participant is instructed to close their eyes and is expected to maintain balance for 30 seconds. The duration of standing on one leg during this time is recorded. If the lifted limb touches the supporting leg, the foot touches the ground, there is swaying or hopping, or if external support is used, it is considered a balance disturbance.
Change in quadriceps femoris muscle thickness after a 6-week exercise program | Baseline and 1 week after the 6-week exercise program
  For the bilateral examination of the muscle thickness of the vastus intermedius and rectus femoris, patients will be positioned in a supine position with knees fully extended. Horizontal imaging will be performed at the midpoint of the line between the anterior superior iliac spine and the upper part of the patella. The average of three measurements will be recorded as the muscle thickness. All measurements will be repeated three times, and the average of these measurements will be used for analysis.
Change in Visual Analog Scale at rest and during activity after a 6-week exercise program | Baseline and 1 week after the 6-week exercise program
  Pain intensity will be evaluated with the Visual Analog Scale (VAS). Patients will be asked about the average pain intensity that they had felt at rest and during activity.
  Therefore, a score closer to 10 reflects a more severe pain experience, while a score of 0 indicates the absence of pain.

CONTACTS AND LOCATIONS:
Overall Officials: İrem Setenay ÖZKAN, Principal Investigator — Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Bahçelievler, Turkey (Türkiye)